CLINICAL TRIAL: NCT01422577
Title: A Randomized Comparison Between White Light Endoscopy (WLE) and Bright Narrow Band Imaging (B-NBI) in the Diagnosis of Colonic Adenomas in Asymptomatic Subjects Undergoing Screening Colonoscopy
Brief Title: Diagnosis of Colonic Adenomas by Bright Narrow Band Imaging (B-NBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B-NBI
Record Dates: First submitted 2011-08-02; First posted 2011-08-24 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Colonic Adenomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright Narrow Band Imaging (Active Comparator): Bright Narrow Band Imaging
  Interventions: Device: Bright Narrow Band Imaging
- White Light Endoscopy (Active Comparator): White Light Endoscopy
  Interventions: Device: White light Endoscopy

INTERVENTIONS:
Device: Bright Narrow Band Imaging — It is a High Definition system with narrow band imaging option in th endoscope.
  Arms: Bright Narrow Band Imaging
Device: White light Endoscopy — White light Endoscopy
  Arms: White Light Endoscopy

SUMMARY:
Early detection of colo-rectal adenoma using colonoscopy can prevent occurrence of colon cancers. While colonoscopy is a standard technique, it can miss early cancers. To improve the detection rate, Narrow Band Imaging (NBI) was introduced in 2006. It has been shown to compare favorably with chromo-endoscopy in the sensitivity and specificity in the diagnosis of malignant colo-rectal neoplasms. The major drawback of NBI is that images become dark in the presence of blood and fecal matters. The bright-NBI is a prototype imaging technology that enables endoscopists to obtain better images in suboptimal conditions. The study proposes to compare the performance of colonoscopy using either white light or bright NBI in subjects undergoing screening colonoscopy in search for colon adenomas.

Purpose

To determine that bright -NBI is superior to WLE in detecting colorectal adenomas in average risk subjects undergoing screening colonoscopy.

DETAILED DESCRIPTION:
Removal of colorectal adenomas prevents occurrence of cancers [1]. It is recognized that colonoscopy can miss colorectal adenomas and early cancers [2]. There is a need to further improve performance of colonoscopy. The use of chromo-endoscopy has been shown to improve detection of flat adenomas [3]. Narrow band imaging was introduced in year 2006. It is similar to chromo-endoscopy in that it provides more mucosal details. This enables endoscopists to accurately describe the pit pattern of adenomas. NBI has been used as a substitute to chromo-endoscopy. In pooled analysis, NBI is comparable to chromo-endoscopy in their sensitivity and specificity in the diagnosis of malignant colorectal adenomas [4]. Unfortunately, the use of NBI has not been shown to conclusively improve rate of colorectal adenoma detection. Two of 3 randomized trials that compared WLE to NBI showed a higher adenoma detection rate with the use of NBI [5, 6]. In a study by Rex et al., the rate was however similar with either modality. In a pooled analysis, NBI was only marginally better than WLE [4].

The effective use of NBI depends on the quality of bowel preparation and the experience of endoscopist. In the presence of fecal matters, NBI tends to be dark and detection of small adenomas becomes difficult. The prototype bright NBI coupled with high definition resolution is likely to overcome this drawback of original NBI.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic subjects undergoing screening colonoscopy
2. age > 40
3. average risk subjects defined as those without a personal history of inflammatory bowel disease, colon adenoma or cancer or family history of Familial adenomatous polyposis (FAP) or Familial non-polyposis syndrome or first degree relatives having diagnosed to have colo-rectal carcinoma
4. no colonoscopy in past 5 years
5. ability to provide a written consent to trial participation

Exclusion Criteria:

1. Patient age < 50
2. Patients with prior colorectal surgery
3. Pregnant or lactating women
4. Colonoscopy done within the past 5 years
5. Lack of consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1006 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Colorectal adenoma detection rate | 2 years
  compare the rate in colorectal adenoma detection between B-NBI and conventional colonoscopy

SECONDARY OUTCOMES:
1. Rate in the detection of advanced neoplasms (defined by adenomas >10 mm in size, with high grade dysplasia or with >25% villous features). | 2 years
  compare the advanced neoplasm detection rate
2. Sensitivity and specificity of either image modality in the diagnosis of malignant adenomas using pathology | 2 years
  compare the sensitivity and specificity between B-NBI and conventional colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: James YW LAU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China